CLINICAL TRIAL: NCT05699577
Title: Prognostic Value of Some Biochemical Markers in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amany Fathy Abdelrasoul, demonestrator at medical biochemistry, Sohag University
Other Study IDs: Soh-Med-23-01-07
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- metastatic breast cancer
  Interventions: Diagnostic Test: serum sample for ELIZA
- non metastatic breast cancer
  Interventions: Diagnostic Test: serum sample for ELIZA

INTERVENTIONS:
Diagnostic Test: serum sample for ELIZA — ELIZA for Ca15-3 and interferon gamma

SUMMARY:
breast cancer is the most common type of cancer in women and first cause of cancer death among them. in Egypt it constitutes 33% of female cancer cases and more than22000 new cases diagnosed each year. there are many prognostic factors for breast cancer as Tumer size, axillary lymph node status, hormonal receptor status, and tumer markers as Ca15-3 and interferon gamma.

ELIGIBILITY:
Inclusion Criteria:

* female patients aged more than or equal 18 year diagnosed with breast cancer
* metastatic and non-metastatic cancer premenopausal and postmenopausal female positive and negative hormonal receptors and HER2 receptor taking any systemic treatment taking radiotherapy or not

Exclusion Criteria:

* female patients less than 18 years patients having comorbid disease. patients with double malignancy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: female patients with breast cancer
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
serum level of Ca15-3 | 6 months
  Tumer marker
serum level of interferon gamma | 6 months
  Tumer marker

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Uygur MM, Gumus M. The utility of serum tumor markers CEA and CA 15-3 for breast cancer prognosis and their association with clinicopathological parameters. Cancer Treat Res Commun. 2021;28:100402. doi: 10.1016/j.ctarc.2021.100402. Epub 2021 May 24. PMID 34082362
- [Background] Jorgovanovic D, Song M, Wang L, Zhang Y. Roles of IFN-gamma in tumor progression and regression: a review. Biomark Res. 2020 Sep 29;8:49. doi: 10.1186/s40364-020-00228-x. eCollection 2020. PMID 33005420
- [Background] Mendoza JL, Escalante NK, Jude KM, Sotolongo Bellon J, Su L, Horton TM, Tsutsumi N, Berardinelli SJ, Haltiwanger RS, Piehler J, Engleman EG, Garcia KC. Structure of the IFNgamma receptor complex guides design of biased agonists. Nature. 2019 Mar;567(7746):56-60. doi: 10.1038/s41586-019-0988-7. Epub 2019 Feb 27. PMID 30814731